CLINICAL TRIAL: NCT06459791
Title: Efficacy of Personalized Tumorogram-based Therapy in Cancer Established From Patient-derived Biological Avatar: Proof-of-concept Study
Brief Title: Efficacy of Personalized Tumorogram-based Therapy in Cancer Established From Patient-derived Organoid (AVATAR)
Acronym: AVATAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC 2023-08
Record Dates: First submitted 2024-05-27; First posted 2024-06-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer
Keywords: tumorogram; metastatic breast cancer; avatar; Organoid; PDO
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy

STUDY DESIGN:
Intervention Model Description: Methodology: RIPH 1, Phase II, multi-center, single-arm, non-randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Line N in step 1 (Other): Step 1: follow-up of line N (standard care) when the tumorogram is established. Intervention is the biopsy performed before start of treatment in line N. Standard of Care treatment
  Interventions: Procedure: Biopsy
- Line N+1 in step 2 (Experimental): Step 2: in case of informative tumorogram: follow-up of experimental line N+1. If tumorogram is informative on organoid issued from biospy, a specific standard of Care treatment will be recommanded.
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — The recommandation done based on informative tumorogram is up to study investigator
  Other Names: Line N+1 treatment recommandation

SUMMARY:
A biopsy of a tumor lesion (breast or other localisation) will be performed for processing to establish avatars (patient-derived organoids -PDO). A personalized tumorogram for each patient will be provided, based on the results of the drug screening (= tumor predicted as sensitive, intermediate, resistant or non-evaluable for each drug tested). Patients with an informative tumorogram will receive one of the recommended treatments (line N+1) in the event of tumor progression, administered according to standard procedures and validated at medical meetings specific to each center, and their fate will be monitored.

DETAILED DESCRIPTION:
A biopsy of a tumor lesion (breast or other localisation) will be performed and transferred to the LIP laboratory at the Institut Curie (Laboratoire d'Investigation Préclinique, Département de Recherche Translationnelle) for processing to establish avatars (patient-derived organoids -PDO).

Step 1: Establishment of avatar (PDO): follow-up of line N (standard care) when the tumorogram is established, then follow-up of standard line N+1.

* The patient will then be treated (line N) as part of standard care while awaiting the result of the tumorogram.
* A drug screening will be carried out on the PDO (~5-10 drugs/patient), which will be progressive and adapted to the clinical context (including treatment history), including drugs used in standard care (cf. list in Table 1).
* A personalized tumorogram for each patient will be provided, based on the results of the drug screening (= tumor predicted as sensitive, intermediate, resistant or non-evaluable for each drug tested).
* A multidisciplinary committee will be set up for this study, which will meet regularly (~1 time per week) to discuss patients included in the study, obtaining PDOs, drugs to be prioritized in the screening, results of the drug screening and personalized tumorograms. The committee will include at least one oncologist and one biologist from the laboratory.
* The multidisciplinary committee will make a therapeutic recommendation based on the personalized tumorogram, which may include several drugs considered sensitive to the tumour
* A tumorogram will be considered as informative if it proposes at least one chemotherapy molecule considered as sensitive in the PDO model.
* Patients whose PDO could not be obtained, or whose tumorogram was not informative, will receive standard treatment.

Step 2: informative tumorogram: follow-up of experimental line N+1 Patients with an informative tumorogram will receive one of the recommended treatments (line N+1) in the event of tumor progression, administered according to standard procedures and validated at medical meetings specific to each center, and their fate will be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Patient over 18 years of age
2. Advanced breast cancer
3. Triple-negative phenotype (HR-/HER2-) or HR+/HER2- after hormone resistance (progression after treatment with hormone therapy + CDK4/6 inhibitor)
4. Tumor measurable according to RECISTv1.1 criteria, accessible to biopsy
5. Performans Status 0-1

Exclusion Criteria:

1. More than 3 lines of chemotherapy in the advanced setting (excluding hormone therapy/CDK4/6 inhibitor)
2. Progressive brain metastases
3. Leptomeningeal metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Tumor response rate | 6 months
  Evaluation in the cohort of patients treated according to the informative tumorogram: tumor response rate within 6 months of the start of this treatment.
  Tumor response is defined as partial or complete response, assessed based on radiological criteria (RECIST v1.1) or clinical criteria where applicable.

SECONDARY OUTCOMES:
Comparison of response rate between both the arms | 6 months
  Comparison of response rate and PFSn+1 (recommended treatment) with response rate and PFSn+1 of patients who did not have an established tumorogram;
Organoid cultures achievement | 6 months
  Percentage of achievement of a PDO
Tumorograms performance | 6 months
  Percentage of informative tumorograms versus number of tumorograms returned
Overall survival | up to 18 months
  Comparison of overall survival (OSn+1, defined as the time between the start of treatment on line n+1 and death) between patients treated according to the tumorogram and patients without a tumorogram and treated according to the guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Luc CABEL, MD, Principal Investigator — Institut Curie
Locations (3):
- France (3):
  - Institut Curie, Paris
  - Hôpital Saint-Louis - AP-HP Senopole, Paris
  - Institut Curie, Saint-Cloud

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share de-identified data sets with interested researchers, educators or clinicians. Materials generated under the project will be disseminated in accrodance with Institut Curie policies.
Supporting Information: Study Protocol, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific reserach, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).